CLINICAL TRIAL: NCT01483079
Title: Evaluation of Post-Discharge Growth and Development of Infants Who Received Donor Human Milk Products in the NICU
Brief Title: Post-Discharge Growth of Infants Who Received Donor Human Milk Products in the Neonatal Intensive Care Unit (NICU)
Acronym: NICU
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: H-29522
Record Dates: First submitted 2011-11-09; First posted 2011-12-01 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prematurity
Keywords: donor human milk products; post-discharge; growth; development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Former preterm infants: A cohort of infants less than or equal to 1250 grams birth weight that received donor human milk products in the NICU will be recruited and followed. Some infants recruited will be from a previously studied population of very low birth weight infants receiving donor human milk products in the NICU at Texas Children's Hospital.

SUMMARY:
Human milk feeding is associated with great benefits to the health and development of infants, especially in premature infants. Some mothers are unable or unwilling to provide breast milk to their infant. The use of donor human milk products for very low birth weight infants as an alternative to cow milk has risen dramatically in the past year.

Purpose: To evaluate post-discharge growth and neurodevelopment of infants less than or equal to 1250 grams birth weight receiving an exclusive human milk protein diet.

DETAILED DESCRIPTION:
An exclusive human milk protein diet in infants less than 1250 grams birth weight has been shown to reduce the rate of necrotizing enterocolitis, a devastating intestinal disease in premature infants, by 50%. New guidelines were introduced in 2009 at Texas Children's Hospital to outline the appropriate use of donor human milk products.

First, infants from a previous study will be identified and recruited for this study. Other potential subjects (infants) will be identified by the GCRC nursing staff at Texas Childrens Hospital upon admission to the neonatal intensive care unit (NICU) (Levels 2 and 3) and communicated to the PI and PIs staff.

This study includes three visits:

1. Outpatient visit at 12 to 15 months corrected gestational age- first outpatient visit to obtain baseline anthropometric data, interim medical history, demographic and socioeconomic information, and nutrition history of the child since discharge (formula, human milk, vitamins, and medications), and check hemoglobin and ferritin. Parents will bring their childs labs from the pediatrician or give permission for records to be accessed in Epic if they receive care from Texas Childrens Pediatric Associates. If records are obtained, labs will not be drawn at this visit. Some of the historical information may be obtained via telephone prior to the outpatient visit.
2. Outpatient visit at 18 to 22 months corrected gestational age- second outpatient visit for collection of anthropometric data, interim medical history, demographic and socioeconomic information, nutrition history, routine Neurodevelopmental Evaluation as part of standard follow-up for extremely low birth weight infants (The Bayley Scales of Infant Development II) administered by certified testers (trained professional), and whole body dual energy x-ray absorptiometry (DXA) will be performed. Some of the historical information may be obtained via telephone prior to the outpatient visit. We will also obtain the height and weight of mom and dad at this visit.
3. Outpatient visit at 5 years of age- third outpatient visit for collection of anthropometric data, interim medical history, demographic and socioeconomic information, nutrition history and developmental evaluation as routine for a school age child. Some of the historical information may be obtained via telephone prior to the outpatient visit.

If infants were not originally followed in the H-26923 study, additional data will be collected from the infants chart for the hospitalization in the NICU. Data collected will include: anthropometrics at birth and discharge, enteral feeding data and parenteral nutrition throughout admission, nutrition related labs, APGAR scores, medications- lasix, chlorothiazide, dopamine, hydrocortisone and dexamethasone, morbidities such as necrotizing enterocolitis, patent ductus arteriosus, spontaneous intestinal perforation, intraventricular hemorrhage, sepsis, and chronic lung disease.

If infants are re-hospitalized or they receive their primary care from a Texas Childrens Pediatrics Associates Clinic, with the consent of the subjects parents, we would collect information from the chart including: interim anthropometric data, interim medical history, nutrition data and history, and nutrition related labs.

No interventions are part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants (<37 weeks gestation) with a birth weight less than or equal to 1250 grams birth weight that received donor human milk products in the NICU during hospitalization.

Exclusion Criteria:

* Infants with a birth weight greater than 1250 grams.
* Infants transferred from an outside hospital to TCH at greater than one week of age.
* Infants who do not achieve any enteral feeds by 4 weeks of age.
* Infants with major congenital anomalies.
* Infants who die within the first 48 hours of admission to TCH.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of infants less than or equal to 1250 grams birth weight that received donor human milk products in the NICU will be recruited and followed. Some infants recruited will be from a previously studied population of very low birth weight infants receiving donor human milk products in the NICU at Texas Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-discharge growth and neurodevelopment | 12-15 months of age
  Per the protocol procedures, growth and development will be assessed at each study visit.
Post-discharge growth and neurodevelopment | 18-22 months of age
  Per the protocol procedures, growth and development will be assessed at each study visit.
Post-discharge growth and neurodevelopment | 5 years of age
  Per the protocol procedures, growth and development will be assessed at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Hair, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States